CLINICAL TRIAL: NCT05469737
Title: A Phase 2/3, Multicenter, Randomized, Dose Optimization (Part I), Double-blind (Part II) Study to Compare the Efficacy and Safety of Oral Azacitidine (Oral-Aza, ONUREG®) Plus Best Supportive Care (BSC) Versus Placebo Plus BSC in Participants With IPSS-R Low- or Intermediate-risk Myelodysplastic Syndrome (MDS)
Brief Title: A Study to Compare the Efficacy and Safety of Oral Azacitidine Plus Best Supportive Care (BSC) Versus Placebo Plus BSC in Participants With International Prognostic Scoring System Revised (IPSS-R) Low- or Intermediate-risk Myelodysplastic Syndrome (MDS)
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA055-026; U1111-1276-5463 (Other Grant/Funding Number: WHO)
Record Dates: First submitted 2022-07-08; First posted 2022-07-22 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Myelodysplastic Syndromes
Keywords: Anemia; Thrombocytopenia
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia; Thrombocytopenia | interventions — Azacitidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part I - Oral-Aza (Dose 1) (Experimental)
  Interventions: Drug: Oral Azacitidine
- Part I - Oral-Aza (Dose 2) (Experimental)
  Interventions: Drug: Oral Azacitidine
- Part II - Oral-Aza (RP3D) (Experimental): RP3D: Recommended Phase 3 Dose
  Interventions: Drug: Oral Azacitidine
- Part II - Placebo (Experimental)
  Interventions: Drug: Placebo for Oral Azacitidine

INTERVENTIONS:
Drug: Oral Azacitidine — Specified dose on specified days
  Other Names: BMS-986345; Oral-Aza; ONUREG®
  Arms: Part I - Oral-Aza (Dose 1); Part I - Oral-Aza (Dose 2); Part II - Oral-Aza (RP3D)
Drug: Placebo for Oral Azacitidine — Specified dose on specified days
  Arms: Part II - Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of oral azacitidine in participants with low to intermediate International Prognostic Scoring System Revised (IPSS-R) myelodysplastic syndrome (MDS).

ELIGIBILITY:
Inclusion Criteria:

• Participant has a documented diagnosis of MDS according to WHO 2016 classification that meets International Prognostic Scoring System Revised (IPSS-R) classification of low- or intermediate-risk disease (IPSS-R score between 1.5 and 4.5).

MDS diagnosis, WHO classification, and IPSS-R risk classification will be prospectively determined by independent central pathology and cytogenetics review, and applicable central laboratory results.

• Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.

Exclusion Criteria:

* Participants with prior malignancies must have an expected median life expectancy of at least 12 months at the time of inclusion and no active treatment of any sort for at least 24 weeks prior to randomization (including but not limited to immunotherapy or targeted therapy)
* Hypoplastic Myelodysplastic Syndrome (MDS) with a marrow cellularity of ≤ 10%
* Participants diagnosed with MDS with excess blasts-2 (MDS-EB2)
* Prior treatment with azacitidine (any formulation), decitabine, or other hypomethylating agent

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-29 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) criteria v.5.0 | 6 cycles plus 28 days (up to 24 weeks)
  Phase 2
Number of participants who achieved complete remission (CR) per International Working Group (IWG) 2006 criteria within 6 cycles | Up to 24 weeks
  Phase 2 and 3

SECONDARY OUTCOMES:
Number of participants who achieved Overall Response (OR) per IWG 2006 criteria within 6 cycles | Up to 24 weeks
  Phase 2 and Phase 3
  Overall Response is defined as complete response (CR), partial remission (PR), marrow complete response (mCR), hematologic improvement-erythroid response (HI-E), hematologic improvement-platelet response (HI-P), or hematologic improvement-neutrophil response (HI-N) as per IWG 2006 criteria
Number of participants who achieved 84-day packed red blood cells transfusion independence (pRBC-TI) | Up to 32 weeks
  Phase 2 and Phase 3
pRBC-TI duration | Over the course of the study, an average of 1 year
  Phase 2 and Phase 3
Number of participants who achieve 84 day platelet transfusion independence (PLT-TI) within 6 cycles | Over the course of the study, an average of 1 year
  Phase 2 and Phase 3
PLT-TI duration | Over the course of the study, an average of 1 year
  Phase 2 and Phase 3
Number of participants who achieved pRBC transfusion reduction | Over the course of the study, an average of 1 year
  Phase 3
pRBC transfusion reduction duration | Over the course of the study, an average of 1 year
  Phase 3
CR duration | Over the course of the study, an average of 1 year
  Phase 2 and Phase 3
Best OR | Over the course of the study, an average of 1 year
  Phase 2 and Phase 3
OR duration | Over the course of the study, an average of 1 year
  Phase 2 and Phase 3
Overall Survival (OS) | Up to 5 years after discontinuation of Investigational Product, approximately 6 years
  Phase 3
Event-free Survival (EFS) | Up to 5 years after discontinuation of Investigational Product, approximately 6 years
  Phase 3
Time to acute myeloid leukemia (AML) | Up to 5 years after discontinuation of Investigational Product, approximately 6 years
  Phase 3
Time to subsequent therapy | Up to 5 years after discontinuation of Investigational Product, approximately 6 years
  Phase 3
Iron parameters measured from blood | Over the course of the study, an average of 1 year
  Phase 3
Number of participants with Adverse Events (AEs) evaluated using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) criteria v.5.0 | Up to end of treatment/early termination, an average of 1 year
  Phase 3
Summary statistics for Functional Assessment of Cancer Therapy-Anemia (FACT-An) scales and subscales at each assessment point for each treatment arm | Up to end of treatment/early termination, an average of 1 year
  Phase 3
Summary statistics for Quality of Life in Myelodysplasia Scale (QUALMS) scales and subscales at each assessment point for each treatment arm | Up to end of treatment/early termination, an average of 1 year
  Phase 3
Summary statistics for the EuroQol 5 Dimension 5 Level (EQ-5D-5L) scales and subscales at each assessment point for each treatment arm | Up to end of treatment/early termination, an average of 1 year
  Phase 3
Number of participants with healthcare resource use associated with the investigational product (IP) | Over the course of the study, an average of 1 year
  Phase 3

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (65):
- United States (7):
  - Local Institution - 0137, Miami, Florida
  - Local Institution - 0147, Tamarac, Florida
  - Local Institution - 0132, East Syracuse, New York
  - Local Institution - 0073, Pittsburgh, Pennsylvania
  - Local Institution - 0014, Houston, Texas
  - Local Institution - 0086, Houston, Texas
  - Local Institution - 0123, Fairfax, Virginia
- Argentina (5):
  - Local Institution - 0070, Pilar, Buenos Aires
  - Local Institution - 0039, ABB, Buenos Aires F.D.
  - Local Institution - 0016, Buenos Aires
  - Local Institution - 0022, Buenos Aires
  - Local Institution - 0050, Buenos Aires
- Australia (4):
  - Local Institution - 0006, Clayton, Victoria
  - Local Institution - 0018, Melbourne, Victoria
  - Local Institution - 0004, Melbourne, Victoria
  - Local Institution - 0003, Melbourne
- Canada (3):
  - Local Institution - 0008, Toronto, Ontario
  - Local Institution - 0015, Toronto, Ontario
  - Local Institution - 0090, Montreal, Quebec
- Local Institution - 0156, Wuhan, Hubei, China
- Local Institution - 0060, Hradec Králové, Czechia
- Denmark (2):
  - Local Institution - 0115, Aarhus, Central Jutland
  - Local Institution - 0116, Aalborg, North Denmark
- France (6):
  - Local Institution - 0063, Pessac, Aquitaine
  - Local Institution - 0024, Tours, Indre-et-Loire
  - Local Institution - 0094, Angers, Maine-et-Loire
  - Local Institution - 0056, Lille, Nord
  - Local Institution - 0085, Villejuif, Val-de-Marne
  - Local Institution - 0082, Paris
- Germany (6):
  - Local Institution - 0081, Duisburg, North Rhine-Westphalia
  - Local Institution - 0128, Düsseldorf, North Rhine-Westphalia
  - Local Institution - 0055, Leipzig, Saxony
  - Local Institution - 0037, Dresden
  - Local Institution - 0007, Hamburg
  - Local Institution - 0028, Mutlangen
- Greece (3):
  - Local Institution - 0125, Chaïdári, Attikí
  - Local Institution - 0129, Thessaloniki, Thessaloníki
  - Local Institution - 0127, Alexandroupoli
- Hong Kong (2):
  - Local Institution - 0178, Hksar
  - Local Institution - 0180, Shatin
- Italy (4):
  - Local Institution - 0061, Rome, Lazio
  - Local Institution - 0052, Rozzano, Milano
  - Local Institution - 0075, Florence, Tuscany
  - Local Institution - 0101, Bologna
- Japan (7):
  - Local Institution - 0136, Kitakyushu-shi, Fukuoka
  - Local Institution - 0154, Sapporo, Hokkaido
  - Local Institution - 0153, Amagasaki, Hyōgo
  - Local Institution - 0130, Sagamihara, Kanagawa
  - Local Institution - 0135, Sendai, Miyagi
  - Local Institution - 0150, Shinagawa-ku, Tokyo
  - Local Institution - 0124, Osaka
- Local Institution - 0097, Olsztyn, Warmian-Masurian Voivodeship, Poland
- South Korea (5):
  - Local Institution - 0058, Hwasun Gun, Jeonranamdo
  - Local Institution - 0048, Seoul, Seoul Teugbyeolsi
  - Local Institution - 0036, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0012, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0051, Junggu, Taegu-Kwangyǒkshi
- Spain (6):
  - Local Institution - 0109, Valencia, Valenciana, Comunitat
  - Local Institution - 0107, Granada
  - Local Institution - 0111, Madrid
  - Local Institution - 0112, Ourense
  - Local Institution - 0110, Oviedo
  - Local Institution - 0108, Salamanca
- Sweden (2):
  - Local Institution - 0118, Stockholm, Stockholms Län [se-01]
  - Local Institution - 0119, Örebro, Örebro Län [se-18]

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05469737.html